CLINICAL TRIAL: NCT03233841
Title: Observational and Cross-Sectional Cohort Study of the Natural History and Phenotypic Spectrum of Farber Disease
Brief Title: Farber Disease Natural History Study
Status: Completed | Type: Observational
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: RVT-801-0001
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Farber Disease; Farber's Disease; Farber Lipogranulomatosis; Acid Ceramidase Deficiency; Ceramidase Deficiency; N-Laurylsphingosine Deacylase Deficiency; ASAH1 Mutation
Keywords: Natural History Study; Observational Study; Prospective Study; Retrospective Study; Farber Disease; Farber's Disease; ASAH1; Subcutaneous Nodules; Lysosomal Storage Disease; Lysosomal Storage Disease, Nervous System; Metabolic Diseases; Lipid Metabolism Disorders; Lipidoses; Sphingolipidoses; Genetic Disease, Inborn; Musculoskeletal Diseases; Connective Tissue Diseases; Central Nervous System Diseases; Brain Diseases, Metabolic, Inborn; Brain Diseases, Metabolic; Brain Diseases, Inborn; Brain Diseases; Infant, Newborn Diseases; Inborn Errors of Metabolism; Inherited Metabolic Disease
MeSH Terms: conditions — Farber Lipogranulomatosis; Lysosomal Storage Diseases; Neurologic Manifestations; Metabolic Diseases; Lipid Metabolism Disorders; Lipidoses; Sphingolipidoses; Genetic Diseases, Inborn; Musculoskeletal Diseases; Connective Tissue Diseases; Central Nervous System Diseases; Brain Diseases, Metabolic, Inborn; Brain Diseases, Metabolic; Brain Diseases; Infant, Newborn, Diseases; Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Living non-HSCT Farber Disease Patients: Patients with a confirmed diagnosis of Farber disease who are currently alive and have not undergone hematopoietic stem cell transplantation (HSCT).
- Living HSCT Farber Disease Patients: Patients with a confirmed diagnosis of Farber disease who are currently alive and have undergone hematopoietic stem cell transplantation (HSCT).
- Deceased Farber Disease Patients: Patients with a confirmed diagnosis of Farber disease who are deceased (including patients who may or may not have undergone hematopoietic stem cell transplantation).

SUMMARY:
The primary objective of this study is to establish the natural history of Farber disease (acid ceramidase deficiency) through the collection and analysis of retrospective and prospective data on patients diagnosed with Farber disease. All patients diagnosed with Farber disease are eligible, including both those who have and have not undergone hematopoietic stem cell transplantation (HSCT). Additionally, data and records from deceased patients will provide valuable retrospective data for this study.

The secondary objective of the study is to establish a set of clinical data, laboratory data (biomarkers), and functional data potentially useful for:

* Assessing the efficacy of HSCT and the efficacy of potential future therapies (for example with RVT-801, recombinant human acid ceramidase) in Farber disease
* Characterizing changes in symptoms of patients over time
* Characterizing distinct groups (phenotypes) within the patient population
* Documenting the disease histories of individual patients to serve as intra-subject control data for those who may enroll in any future clinical studies with therapies for Farber disease

The exploratory objectives of the study are:

* To explore the relationship between patient disease activity or phenotype and specific ceramide levels or specific immunologic markers (cytokines/chemokines) in blood
* To evaluate a standardized tool, the Farber Disease Natural History Instrument (FDNI), to be used for the collection of patient history information, data from clinical, laboratory, genetic, and functional studies, and data from review of medical records

ELIGIBILITY:
Inclusion Criteria:

* Living or deceased subjects with diagnosis of Farber disease, based on clinical (typical clinical symptoms) and biochemical and/or genetic criteria, as follows:

  * Biochemical: An acid ceramidase activity value in white blood cells, cultured skin fibroblasts or other biological sources (e.g., plasma) that is less than 30% of control (normal) values established by the testing laboratory. For deceased subjects only, storage of ceramide in cells from histopathologic sections is also adequate to confirm the diagnosis.
  * Genetic: Nucleotide changes within both alleles of the acid ceramidase gene (ASAH1) or cDNA that indicate, through bioinformatics, gene expression studies, or other methods, a possible loss of function of the acid ceramidase protein.
* Informed consent or assent, for living subjects. For deceased subjects it is the responsibility of the principal investigator to ensure that the proper requirements are met according to local laws and regulations.

Exclusion Criteria:

• Current use or history of use in the past 30 days of an investigational agent (with exception of off-label use of medications).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All identified patients with Farber disease, living or deceased, diagnosed by biochemical or genetic criteria, or both, are eligible for inclusion in the study without regard to any other baseline or demographic characteristics. Both subjects who have undergone HSCT and those who have not are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-10-12 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Establish a dataset on the natural history of Farber Disease | Up to 21 months
  Collection of information for all subjects will include data from:
  * Medical history
  * Farber disease diagnosis, presentation, treatments and symptom progression
  Collection of information from living subjects will include:
  * Medical examination
  * Disease-specific data (Farber Disease Natural History Instrument - FDNI)
  * Laboratory tests (laboratory assessments and inflammatory markers)
  * Functional tests
    * Six-minute walk test (6MWT)
    * Pulmonary function testing
  * Additional assessments and evaluations:
    * Patient reported outcomes
    * Pain assessment
    * Relative impact of symptoms
    * Nodule Impact Questionnaire
    * Physician and Patient/Parent global assessment
    * Measurement and clinical characteristics of index nodules
    * Ultrasound evaluation of liver and spleen
    * High-frequency ultrasound

CONTACTS AND LOCATIONS:
Locations (15):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's National Health System, Washington D.C., District of Columbia
- Hospital de Niños de la Santisima Trinidad, Córdoba, CP, Argentina
- Montreal Children's Hospital, Montreal, Quebec, Canada
- Cairo University, Cairo, Egypt
- Universitätsklinikum Giessen, Zentrum für Kinderheilkunde und Jugendmedizin, Giessen, Hesse, Germany
- India (2):
  - Lok Nayak Hospital & Maulana Azad Medical College, Dehli
  - Sir Ganga Ram Hospital, Delhi
- Italy (2):
  - IRCCS Istituto Giannina Gaslini, Genoa
  - University of Milan, Milan
- Astrid Lindgrens barnsjukhus, Karolinska University Hospital Solna, Stockholm, Sweden
- Turkey (Türkiye) (4):
  - Cukurova University School of Medicine, Adana
  - Hacettepe University Medical Faculty Hospital, Ankara
  - Istanbul University Istanbul School of Medicine, Istanbul
  - Dokuz Eylul University School of Medicine, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elsea SH, Solyom A, Martin K, Harmatz P, Mitchell J, Lampe C, Grant C, Selim L, Mungan NO, Guelbert N, Magnusson B, Sundberg E, Puri R, Kapoor S, Arslan N, DiRocco M, Zaki M, Ozen S, Mahmoud IG, Ehlert K, Hahn A, Gokcay G, Torcoletti M, Ferreira CR. ASAH1 pathogenic variants associated with acid ceramidase deficiency: Farber disease and spinal muscular atrophy with progressive myoclonic epilepsy. Hum Mutat. 2020 Sep;41(9):1469-1487. doi: 10.1002/humu.24056. Epub 2020 Jun 24. PMID 32449975
- See also: Related Info — http://www.enzyvant.com/